CLINICAL TRIAL: NCT05697939
Title: Prospective Validation of 3D Body Surface Modeling for Patient Monitoring in Adolescent Idiopathic Scoliosis
Brief Title: 3D Body Surface Modeling for Scoliosis Monitoring
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kali Tileston, Clinical Assistant Professor, Orthopaedic Surgery, Stanford University
Other Study IDs: 54100
Record Dates: First submitted 2023-01-14; First posted 2023-01-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adolescent Idiopathic Scoliosis: Reproducibility group
  Interventions: Diagnostic Test: NSite 3D Scanning

INTERVENTIONS:
Diagnostic Test: NSite 3D Scanning — Three separate users will enter the exam room and use the NSite application to scan the patient in the bending position. These users may include research coordinators, physicians, or other authorized staff.
  The NSite application will have a user tutorial on how to scan patients that users are instructed to watch prior to conducting a scan.
  All participants are asked to remove clothing above the waist but may keep a bra or tight-fitting shirt on during the scanning procedures. The patient will be asked to assume a forward bending position. One user will capture a scan of the patient's back in this position. The user will calibrate the device and then walk around the patient while scanning per app directions. Once this user captures the scan, it will be processed by the application. New scans will then be obtained by the two other users. Once all users have captured a scan, the scanning process and patient participation will be completed.

SUMMARY:
This is a single center, prospective, non-randomized reproducibility study of the NSite device in patients undergoing evaluation for scoliosis. The NSite device is a pre-market, investigational device. The study will enroll 13 eligible patients, who will be scanned using the NSite device by 3 separate users in order to assess if the device generates similar results across users. This data will be used to support 510(k) submission.

DETAILED DESCRIPTION:
The primary objective of this study is to validate the reproducibility of device output in multiple users in a clinical setting. Device output will be predicted probability of major curve magnitude (i.e., Cobb angle) greater than or equal to 20 degrees with 95% confidence interval. We will test whether users obtain similar device output when measuring the same participant (at least 2 scans required for analysis). After excluding bad quality scans, the measurements obtained by these different users (at least 2 users after excluding bad scans) on each study participant will then be compared to determine if they are congruent (having overlapping confidence intervals) or different. The percentage of participants for which users generated congruent predicted probabilities will be reported.

The NSite Scoliosis Assessment App is intended as a clinical decision support tool and requires interpretation by the healthcare professional. It is intended for use for children and adolescent patients 10 to 18 years old. It is for use by prescription only. The NSite Scoliosis Assessment App provides a calculated Asymmetry Index for patients with or at risk for scoliosis, which will yield an output of percentage risk of major curve magnitude (i.e., Cobb angle) greater than 20 degrees, with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10 and 18 years old
* Referred for evaluation of or diagnosed of adolescent idiopathic scoliosis

Exclusion Criteria:

* Scoliosis caused by another condition (e.g., secondary scoliosis)
* Parents/guardians unable to consent
* English is not the primary language (to avoid miscommunication)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with adolescent idiopathic scoliosis, ages 10-18
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess the reproducibility of NSite device | Anticipated to take about one month in order to recruit, enroll, and scan 13 patients.
  Percentage of scan outputs reproducible. The percentage of scan sets (3 scans for each participant) that have reproducible predicted probabilities for major curve magnitude ≥ 20 degrees. A reproducible output will be defined as a scan set in which all scans have overlapping 95% confidence intervals for the predicted probability of major curve magnitude ≥ 20 degrees.

SECONDARY OUTCOMES:
User Feedback | Anticipated to take about one month in order to recruit, enroll, and scan 13 patients.
  User feedback will be collected throughout testing in the form of open-ended comments. These will be collated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kali Tileston, MD, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No